CLINICAL TRIAL: NCT06231134
Title: The Effect of Diode Laser 940 Nm Versus Electrosurgical Device During Second Stage Implant Surgery on Bone and Soft Tissue Healing (A Randomized Controlled Clinical Trial)
Brief Title: Diode Laser 940 Nm Versus Electrosurgical Device During Second Stage Implant Surgery on Bone and Soft Tissue Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0801-11/2023
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Dental Implant; Bone Healing; Soft Tissue Healing
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional surgery (Active Comparator)
  Interventions: Device: Conventional surgery
- Dioad laser (Experimental)
  Interventions: Device: Diode laser 940 nm
- Electrosuregry (Experimental)
  Interventions: Device: Electrosurgical

INTERVENTIONS:
Device: Conventional surgery — an implant will be exposed using the conventional surgical exposure techniques with a tissue punch, the cover screw will be removed, and the healing abutment placed
  Arms: Conventional surgery
Device: Diode laser 940 nm — implant will be uncovered using a diode laser (940nm) in contact type with a continuous mode at a power of 1.5 watts, the laser tip will be used in a circular motion to create a small opening which will be increased till large enough to expose and remove the cover screw and place the healing abutments.
  Arms: Dioad laser
Device: Electrosurgical — the monopolar electrosurgical device will be used in the same way as the laser tip with additional care avoiding contacting the implants during exposure.
  Arms: Electrosuregry

SUMMARY:
Background: Dental lasers and electrosurgical devices have been introduced a long time ago. However, limited studies are available concerning their use in the second stage of implant surgery, with the conventional surgical technique being the standard of care.

Aim of this study: To evaluate clinically and radiographically soft and hard tissue healing associated with the use of electrosurgical and laser devices and compare them with conventional surgical techniques during second-stage implant surgery.

Plan of the study: A randomized controlled clinical trial. The sample size will include patients who have an implant already placed and ready for second stage surgery recruited from the patient pool at the outpatient clinics.

Materials and Methods: Patients will be randomly allocated into the three groups. In Group (A) implant will be exposed using the conventional surgical exposure techniques with a tissue punch, the cover screw will be removed, and the healing abutment placed. In group (B) implant will be uncovered using a diode laser (940nm) in contact type with a continuous mode at a power of 1.5 watts, the laser tip will be used in a circular motion to create a small opening which will be increased till large enough to expose and remove the cover screw and place the healing abutments. In group (C) the monopolar electrosurgical device will be used in the same way as the laser tip with additional care avoiding contacting the implants during exposure.

The outcome: will be soft tissue healing and crestal marginal bone loss around implants.

Soft tissue healing will be assessed on the operative day, 2 weeks, and 4 weeks using Landry index. Crestal bone loss will be assessed using a standardized periapical x-ray at baseline and after 1 month with periapical x-ray.

ELIGIBILITY:
Inclusion Criteria:

* Adequate zone of keratinized mucosa.
* Osseointegrated Implants ready for second-stage surgery.

Exclusion Criteria:

* Heavy smokers due to increased risk of infection, delayed wound healing, and poor immune response.
* Medically compromised patients due to affection of the peri-implant health and tissue maintenance.
* Bad oral hygiene
* Patients with an exposed cover screw
* Evidence of bone loss in the preoperative peri-apical radiograph.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline and after 1 week
  Pain intensity using a Visual Analogue Scale (VAS) score (0 to 10 cm), with a VAS marker of 0-2.50 cm for mild pain; 2.60-5.00 cm for moderate pain; 5.10-7.50 cm for severe pain; 7.60-10.0 cm for unbearable pain (11) during the operative day and the following 7 days.
Change in soft tissue healing | after 1 and 2 weeks
  Soft tissue healing using the Landry index where the following 4 parameters: tissue color, response to palpation, granulation tissue, and incision margin will be assessed with a 5-level score (1= very poor to 5= Excellent). The healing index will be recorded at 2 and 4 weeks.

SECONDARY OUTCOMES:
Change in creastal bone loss | Baseline and 1 month
  Crestal Bone loss following implant exposure using standardized periapical x-ray with implants platform as a reference, with the use of XCP dental x-ray film holder at baseline and after 1 month then the radiographic subtractive measure will be applied to measure the amount of marginal bone loss

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No